CLINICAL TRIAL: NCT05582200
Title: Selective PET Imaging of Astrocytes and Microglia in Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00030631
Record Dates: First submitted 2022-10-07; First posted 2022-10-17 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease; Healthy
MeSH Terms: conditions — Alzheimer Disease | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy subjects
  Interventions: Diagnostic Test: Positron Emission Tomography (PET) using two PET tracer under IND
- Patients with Alzheimer's disease: Patients with Alzheimer's disease
  Interventions: Diagnostic Test: Positron Emission Tomography (PET) using two PET tracer under IND

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography (PET) using two PET tracer under IND — Positron Emission Tomography

SUMMARY:
Inflammation occurs in many brain diseases including Alzheimer's disease. In Alzheimer's disease, amyloid starts accumulating decades before the start of forgetfulness. Basic scientists have reported that inflammation but not amyloid is linked to forgetfulness. When people pinch a finger, it gets swollen. Similar changes occur in brain from various causes. New medications are under development to help healing and prevent permanent damages in the brain. When people pinch a finger, they can check if the injury is healing or getting worse by watching. Investigators can watch inside of the brain using a special camera called positron emission tomography (PET). It is currently possible to watch inflammation in the brain by taking pictures of a molecule called translocator protein (TSPO). But the problem is that by imaging TSPO, investigators can catch changes in more than one kind of cells. The information is not specific to each cell type. Such vague information is not useful to monitor the effect of new medications for inflammation. This proposal attempts to develop a novel method to capture changes in each of two major players in inflammation, microglia and astrocytes. To do so, investigators will take selective pictures of one cell type by using a novel imaging agent for PET. Investigators will also take PET pictures of TSPO. Investigators will process these two kinds of PET pictures using advanced mathematical methods and extract specific information on microglia and astrocytes. Our novel method will be useful to monitor new therapies to treat inflammation in brain.

DETAILED DESCRIPTION:
Inflammation in brain plays critical roles in disease progress and symptom development in a number of brain disorders such as Alzheimer's disease (AD), traumatic brain injury, major depressive disorder, epilepsy, and schizophrenia. Neuroinflammation has been imaged using positron emission tomography (PET) by using translocator protein (TSPO) as the marker. Although TSPO PET studies have provided insight to understand the pathology, some results are difficult to interpret. TSPO imaging has a major limitation of not being selective to one type of glia; it is expressed by both microglia and astrocyte. The current study attempts to overcome this limitation. Monoamine oxidase type-B (MAO-B) is highly expressed by astrocyte and serotonin (5-HT)-releasing neurons but not by microglia. PET studies using a prototype tracer 11C-L-deprenyl detects astrogliosis in mild cognitive impairment (MCI) but this tracer has low levels of specific binding. Preliminary results show that a novel tracer 18F-SMBT-1 developed by Dr. Okamura and his colleagues has several times greater levels of specific binding. The Aims of the current study are to 1) estimate radiation-absorbed doses in 8 healthy people, 2) measure ratios of specific-to-nondisplaceable binding by performing brain scans with and without binding blockade in 5 patients with Alzheimer's disease, 3) measure reproducibility of measuring 18F-SMBT-1 in 8 healthy people, 4) compare MAO-B levels between healthy controls (n = 25) and patients with AD (n = 25), and 5) from 11C-ER176 for TSPO and 18F-SMBT-1, extract cell type specific information for microglia and astrocytes and investigate changes in each cell type In AD.

ELIGIBILITY:
Patients with Alzheimer's disease

Inclusion criteria:

* Individuals of either sex, 50-90 years of age.
* Meeting research criteria for AD (McKhann, Knopman et al. 2011).
* With a CDR (Morris 1993) score of 1-3.
* Fluent in English or Spanish.
* Have sufficient communication and comprehension ability to consent to the performance of the study or have a legally authorized representative.

Exclusion criteria:

* Inability to undergo MRI or PET for any reason, including severe claustrophobia.
* History of large stroke or brain trauma, multiple sclerosis or other brain disorder that, in the judgment of the PI may confound the study.
* Pregnancy. In women in whom the possibility of pregnancy cannot be excluded, a pregnancy test must be performed on site the morning of any PET visit and a negative result together with a physician interview are required prior to the administration or any radiopharmaceutical.
* Research radiation exposure greater than 50 mSv effective dose within 12 months including radiation exposure from this study.

Healthy volunteers:

Inclusion criteria:

* Individuals of 18-90 years of age.
* Negative amyloid accumulation determined by PET (only for the comparison with AD).
* Fluent in English.
* Have enough communication and comprehension ability to consent to the performance of the study.

Exclusion criteria:

* Inability to undergo MRI or PET for any reason, including severe claustrophobia.
* Brain disorder, other than idiopathic headache.
* Current primary Axis I or II psychiatric disorder.
* Current use of psychotropic or anti-epileptic medication.
* Substance abuse during the past two years.
* Active cancer, metabolic encephalopathy, infection, cardiovascular disease.
* Active hematological, renal, pulmonary, endocrine or hepatic disorders, except for treated thyroid disease.
* Pregnancy. In women in whom the possibility of pregnancy cannot be excluded, a pregnancy test must be performed on site the morning of any PET visit and a negative result together with a physician interview are required prior to the administration or any radiopharmaceutical
* Research radiation exposure greater than 50 mSv effective dose within 12 months including radiation exposure from this study.
* Only for the subjects undergoing the blocked scan with selegiline: known contraindications to selegiline, including hypersensitivity to the drug and use of opioids, such as meperidine and some antidepressants such as bupropion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The level of monoamine oxidase-B | At the time of the PET scan
  Binding of PET tracer [F-18]SMBT-1 to monoamine oxidase-B
The level of translocator protein | At the time of the PET scan
  Binding of PET tracer [C-11]ER176 to translocator protein

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States